CLINICAL TRIAL: NCT04547920
Title: A Prospective Efficacy Study Comparing FREquency of Use and Efficacy of a Personalized Surgery-free Wearable and Personalized Bladder Modulation System With Objective Confirmation of Nerve Activation for Use in the Home by Subjects With OverActive Bladder Syndrome
Brief Title: FREEOAB Study for Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avation Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMHOAB2001
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Overactive Bladder; Urinary Frequency; Urinary Incontinence, Urge; Urinary Urgency
Keywords: Neuromodulation; Closed-Loop Neuromodulation; Wearable Neuromodulation; Tibial Nerve Stimulation; Continuous Sensing; Automatic Adjustment
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 12 Weeks Followed by Optional 12 Month Continuation (Experimental): Initial 12 Weeks: Patients were instructed to therapy using a wearable closed-loop, continuous sensing tibial nerve stimulation.
  Optional Months 4-12: Subjects who qualified for the long-term follow up and elected to enroll, signed a new informed consent and continued therapy sessions for the duration of the trial.
  Interventions: Device: Wearable Bladder Modulation System

INTERVENTIONS:
Device: Wearable Bladder Modulation System — Wearable Closed-Loop, Continuous Sensing Tibial Nerve Stimulation Device

SUMMARY:
This is a prospective, multicenter study that was conducted to evaluate the safety and efficacy of a novel, closed-loop, continuous-sensing wearable neuromodulation system for Overactive Bladder symptom control.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and 18 years of age or older at the time of enrollment
2. Willing and capable of giving informed consent
3. Willing and able to comply with study-related requirements and procedures
4. Are an appropriate candidate for the system required in this study based on the clinical judgment of the Investigator.
5. Have been diagnosed or have symptoms of OAB for at least 3 months Page 8 of 30 Version 1.0 dated July 06, 2020 prior to enrollment
6. Have an average of 10 or more frequency events per day in a 3-Day Voiding Diary
7. Able to provide clear, thoughtful responses to questions and questionnaires
8. Able to toilet self and have and maintain personal hygiene
9. Able to don and doff the bladder modulation garment on their ankle area, replace Gel Pads and use the controller
10. Have ankle and foot anatomy that allows the garment to fit properly, including having the hook and loop closures close and without excessive gapping and allowing the electrodes to fit firmly on the skin.
11. Able to sense and tolerate stimulation for the entire 30-minute therapy session
12. Has detectable EMG signal in response to modulation system stimulation during an investigator supervised screening session
13. If currently on medications that may affect their OAB symptoms, is on a stable dose (no new, discontinued, or change in dose) of all prescribed medication for at least 4 weeks prior to enrollment
14. Female subjects of child-bearing potential must have a negative urine dip stick pregnancy test at baseline
15. Have access to Wi-Fi at least weekly
16. Are capable of using the tablet-based controlling app

Exclusion Criteria:

1. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcomes, in the opinion of the investigator.
2. Allergic, or have shown hypersensitivity, to any materials of the system which come into contact with the body
3. Have a pacemaker or implanted defibrillator
4. Have a documented current or reoccurring Urinary Tract Infection (3 or more in the 12months prior to enrollment)
5. Current use of a marketed device for treatment of their OAB or incontinence (including but not limited to Interstim®)
6. Have had Botox treatment for their OAB in the previous 8 months
7. Current use of transcutaneous electric nerve stimulation (TENS) in pelvic region, back or legs
8. Had PTNS treatment within 6 months prior to enrollment
9. Use of investigational drug/device therapy within past 12 weeks
10. Is concomitantly participating in another clinical study
11. Had within 6 months of enrollment a significant untreated substance abuse disorder or polysubstance abuse disorder stemming from dependency producing medications, alcohol, and/or illicit drugs
12. Pregnant or planning to become pregnant within the next 12 weeks
13. Has scar tissue, metal, or other implant in the target ankle that would interfere with stimulation
14. Has a neurological disorder that causes abnormal sensations in the lower leg (loss of sensation or allodynia)
15. Has a neurological disorder that affects the bladder or a diagnosis of interstitial cystitis, radiation cystitis, or fistulas.
16. Has a skin condition in the area of the ankle stimulation location that would preclude them from using surface stimulation
17. Has been diagnosed with incontinence due to neurogenic bladder
18. Have failed a third line treatment for their OAB because of lack of effectiveness in the last 2 years (PTNS, Botox, or SNS)
19. Urge incontinence due to stress predominant mixed urinary incontinence (greater that 60% of the time)
20. Have polyuria (>2500 cc urine output per day)
21. Has urinary retention or incomplete bladder emptying
22. Has symptoms of benign prostatic hyperplasia (BPH -weak stream, straining, hesitancy or intermittency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Stanford University, Stanford, California
  - The Pelvic Solutions Center, Denver, Colorado
  - Colorado Pelvic Floor Consultants, Englewood, Colorado
  - Women's Health Institute, Oak Lawn, Illinois
  - Urology of Indiana, Greenwood, Indiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Michigan Institute of Urology, Saint Clair Shores, Michigan
  - Tranquil Medical Rsearch, Webster, Texas
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 12 Weeks Followed by Optional 12 Month Continuation: Initial 12 Weeks: Patients were instructed to complete therapy with a wearable closed-loop, continuous sensing tibial nerve stimulation device for bladder modulation.
  Optional Months 4-12: Subjects who qualified for the long-term follow up and elected to enroll, signed a new informed consent and continued therapy for the duration of the study.
Period: Initial 12-Week Study
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Started | 96
Completed | 88
Not Completed | 8
Period: Optional 12-Month Long Term Follow-Up
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Started (The Long Term Follow-Up portion of the trial was optional so not every subject who completed the 12-Week portion opted to enter into this portion of the trial.) | 50
Completed | 39
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 84
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White / Caucasian | 77
  Black / African American | 10
  Asian | 3
  Other | 6
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 164 (9.11)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 83.7 (26.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders in Voiding (Urinary Frequency) Events
Description: The percentage of responders in voiding (urinary frequency) events, where a responder is defined as a subject that either achieves a 50% or greater reduction, from baseline (Visit 1) to Week 12 (Visit 5), in total voids per day relative to an upper normal limit of 8 voids per day, or returns to normal (8 or fewer voids per day) at Week 12.
Time Frame: 12 Weeks
Population: Number of Subjects with Reported Voiding Symptom (Avg > 8 / day) at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Number analyzed (Participants) | 89
Participants | 55

2. Secondary Outcome: Percentage of Responders in Incontinence (Leak) Events (IE)
Description: Percentage of Responders in Incontinence (Leak) Events (IE), where a responder is defined as a subject that either achieves a 50% or greater reduction, from baseline (Visit 1) to Week 12 (Visit 5), in total incontinence events per day, or returns to normal (0 events per day), at Week 12.
Time Frame: 12 Weeks
Population: Number of Subjects with Reported Urgency Symptom (Avg Daily Urges > 0) at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Number analyzed (Participants) | 76
Participants | 47

3. Secondary Outcome: Percentage of Responders in Urgency Events (UE)
Description: Percentage of Responders in Urgency Events (UE), where a responder is defined as a subject that either achieves a 50% or greater reduction, from baseline (Visit 1) to Week 12 (Visit 5), in total urgency events per day, or returns to normal (0 events per day) at Week 12.
Time Frame: 12 Weeks
Population: Number of Subjects with Reported Incontinence Symptom (Avg Daily Leaks > 0) at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Number analyzed (Participants) | 74
Participants | 41

4. Secondary Outcome: Overall Responder Rate at 12 Weeks
Description: Overall Responder Rate at 12 Weeks, where responder is defined as any subject with a 50% or greater improvement, or return to normal, in the total number of voids per day, or the total number of urgency events/day, or the total number of leaks per day from baseline at Week 12.
Time Frame: 12 Weeks
Population: Number of Subjects with ≥ 50% Change in Any Symptom
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Number analyzed (Participants) | 94
Participants | 74

5. Secondary Outcome: Overall Responder Rate at 12 Months
Description: Overall Responder Rate at 12 Months, where responder is defined as any subject with a 50% or greater improvement, or return to normal, in the total number of voids per day, or the total number of urgency events/day, or the total number of leaks per day from baseline at 6 months.
Time Frame: 12 Months
Population: # of Subjects with ≥ 50% Change in Any Symptom
Measure: Count of Participants; unit: Participants
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
Number analyzed (Participants) | 39
Participants | 30

ADVERSE EVENTS:
Time Frame: Length of Study (12 months)
Arm/Group | 12 Weeks Followed by Optional 12 Month Continuation
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 17/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 Weeks Followed by Optional 12 Month Continuation (N=96)
Pollakiuria (Frequent Urination) (Renal and urinary disorders) | 4
Foot Pain / Intense Stimulation (Musculoskeletal and connective tissue disorders) | 3
Muscle Spasm (Foot Cramping) (Musculoskeletal and connective tissue disorders) | 2
Foot Contusion (Skin and subcutaneous tissue disorders) | 1
Paraesthesia (Tingling Sensation) (Nervous system disorders) | 2
Thermal Burn (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 2
Varicose Veins (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Potential limitations exist in the inherent design of the trial with use of patient-reported outcomes. This trial also had no control arm and relied on placebo rates available in the published literature. The end points were refined based on FDA feedback and the data was analyzed post-hoc. The opt-in process for the long-term follow-up population may have skewed in favor of patients with better outcomes during Phase I of the study and led to low number of subjects who entered Phase II.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT04547920/Prot_SAP_001.pdf